CLINICAL TRIAL: NCT00672347
Title: Comparison of Clonidine and Morphine Plus Bupivacaine in Caudal Peridural Anesthesia for Postoperative Analgesia After Pediatric Urogenital Surgery
Brief Title: Clonidine and Morphine in Caudal Anesthesia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Santa Casa de Misericórdia de Belo Horizonte (Other)
Responsible Party: Renato Santiago Gomez - PhD,MD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 210665
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Postoperative Pain
Keywords: caudal anesthesia, clonidine, morphine, bupivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Clonidine; Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- B (Active Comparator): compare caudal anesthesia with bupivacaine alone or in addition to morphine, clonidine or both
  Interventions: Drug: Bupivacaine
- C (Active Comparator): compare caudal anesthesia with bupivacaine plus clonidine with caudal anesthesia with bupivacaine alone or in addition to morphine or morphine plus clonidine
  Interventions: Drug: Clonidine
- M (Active Comparator): compare caudal anesthesia with bupivacaine plus morphine with caudal anesthesia with bupivacaine alone or in addition to clonidine or morphine plus clonidine
  Interventions: Drug: Morphine
- CM (Active Comparator): compares caudal anesthesia with bupivacaine, morphine and clonidine with caudal anesthesia with bupivacaine alone or in addition to morphine or clonidine
  Interventions: Drug: Bupivacaine plus clonidine and morphine

INTERVENTIONS:
Drug: Clonidine — 1 mcg/kg
  Arms: C
Drug: Morphine — 20 mcg/kg
  Arms: M
Drug: Bupivacaine plus clonidine and morphine — bupivacaine 0,166% 1 ml/kg
  clonidine 1 mcg/kg
  morphine 20 mcg/kg
  Arms: CM
Drug: Bupivacaine — Caudal anesthesia with bupivacaine 0,166% 1 ml/kg
  Arms: B

SUMMARY:
Hypothesis: The combined use of Clonidine and Morphine in caudal anesthesia provides better postoperative analgesia than either drug alone after urogenital pediatric surgery.

DETAILED DESCRIPTION:
It is a randomized, double blind study, involving 80 children with ages from 1 to 10 years old, submitted to urogenital surgery, under general anesthesia and caudal block. The patients will be divided into 4 groups: bupivacaine alone, bupivacaine plus clonidine, bupivacaine plus morphine, bupivacaine plus clonidine and morphine. The peroperative consumption of analgesics and inhaled gases, BIS, heart rate and arterial blood pressure will be recorded. Postoperative pain will be evaluated by using Wong-Baker faces scale and pain and discomfort score scale, as well as the consumption of analgesics.

ELIGIBILITY:
Inclusion Criteria:

* Urogenital pediatric surgery
* Status physical(ASA) 1 and 2

Exclusion Criteria:

* Cutaneous infection in puncture site

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The overall postoperative consumption of analgesics. | 24 hours

SECONDARY OUTCOMES:
The peroperative consumption of volatile anesthetics. | 3 hours
The peroperative Bispectral Index measure. | 3 hours
Postoperative Wong-Baker faces scale | 24 hours
Postoperative pain and discomfort score scale | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Renato S Gomez, PhD, MD, Study Director — Federal University of Minas Gerais; Magda L Fernandes, M, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Santa Casa de Belo Horizonte Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Tripi PA, Palmer JS, Thomas S, Elder JS. Clonidine increases duration of bupivacaine caudal analgesia for ureteroneocystostomy: a double-blind prospective trial. J Urol. 2005 Sep;174(3):1081-3. doi: 10.1097/01.ju.0000169138.90628.b9. PMID 16094063
- [Background] Luz G, Innerhofer P, Oswald E, Salner E, Hager J, Sparr H. Comparison of clonidine 1 microgram kg-1 with morphine 30 micrograms kg-1 for post-operative caudal analgesia in children. Eur J Anaesthesiol. 1999 Jan;16(1):42-6. doi: 10.1046/j.1365-2346.1999.00430.x. PMID 10084100
- [Background] Vetter TR, Carvallo D, Johnson JL, Mazurek MS, Presson RG Jr. A comparison of single-dose caudal clonidine, morphine, or hydromorphone combined with ropivacaine in pediatric patients undergoing ureteral reimplantation. Anesth Analg. 2007 Jun;104(6):1356-63, table of contents. doi: 10.1213/01.ane.0000261521.52562.de. PMID 17513626